CLINICAL TRIAL: NCT06892639
Title: Evaluation of Dabocemagene Autoficel (D-Fi; FCX-007; Genetically Modified Autologous Human Dermal Fibroblasts) for the Treatment of Wounds Due to Dystropic Epidermolysis Bullosa
Brief Title: Evaluation of D-Fi for the Treatment of Wounds Due to DEB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCB-EB-304
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: DEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: Intra-patient Randomized and Controlled, Open-label, Rater-Blinded, Multi-center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- D-Fi COL7A1 Genetically-Corrected Autologous Fibroblasts (Experimental): Intra-subject randomized (paired wounds in each subject receive experimental treatment, D-Fi, or remain untreated). One target wound pair will be identified for each subject. Following pairing, target wounds will be randomly assigned as the treatment wound (D-Fi is administered) or control wound. Subjects will receive intradermal injections of D-Fi in each specified treatment wound in two or more treatment sessions. The first treatment session occurs at Day 1, the second at Week 8/Month 2 and the third at Week 16/Month 4. Additional treatment sessions may occur at Week 26/Month 6, Week 32/Month 8 and Week 40/Month 10 when unclosed treatment wounds may be re-treated, and unclosed control wounds may be treated.
  Interventions: Biological: D-Fi

INTERVENTIONS:
Biological: D-Fi — D-Fi is composed of fibroblasts isolated from the subject's skin biopsies which are genetically corrected with the full length COL7A1 gene encoding for type VII collagen.

SUMMARY:
The purpose of this study is to determine whether administration of D-Fi in addition to standard of care improves wound healing as compared to standard of care alone (control) in children, adolescents, and adults with Dystrophic Epidermolysis Bullosa.

DETAILED DESCRIPTION:
CCB-EB-304 is a multi-center, intra-patient randomized and controlled, open-label, rater-blinded Phase 3 study of D-Fi for the treatment of persistent non-healing and recurrent DEB wounds in approximately 32 subjects. Each subject will serve as his/her own control. Each subject's Target Wounds will be paired then randomized to receive D-Fi (Treatment Wound) or remain untreated (Control Wound). One Target Wound Pair will be identified for each subject.

Subjects will receive intradermal injections of D-Fi in each specified Treatment Wound in three or more treatment sessions. The first treatment session occurs at Day 1, the second at Week 8/Month 2 and the third at Week 16/Month 4. Additional treatment sessions may occur at Week 26/Month 6 and Week 32/Month 8 and Week 40/Month 10 when unclosed Treatment Wounds may be re-treated, and unclosed Control Wounds may be treated. Safety and efficacy assessments will occur at scheduled intervals through Week 48/Month 12, when the Treatment Period is completed, and is followed by an optional Open-Label Extension (OLE) treatment phase of an additional 96 weeks. A long-term safety follow-up period (through 15 years) commences for subjects who have received one or more D-Fi injections, either following the treatment phase or if the subject had opted-in, the OLE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥2 years of age at the Screening visit
* Clinical diagnosis of DEB with confirmation of COL7A1 genetic mutation.

Exclusion Criteria:

* Medical instability limiting ability to travel to the investigative site.
* Active infection with human immunodeficiency virus, hepatitis B or hepatitis C.
* The presence of clinically significant COL7 antibodies.
* Evidence of systemic infection.
* Known allergy to any of the constituents of the product.
* Female who is pregnant or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2042-02 (Estimated)

PRIMARY OUTCOMES:
The difference in Complete (100%) Wound Closure of the Target Wound Pair at either Week 22 (Visit 6), and Week 24 (Visit 7) or at Week 24 (Visit 7) and Week 26 (Visit 8) as assessed by a Blinded Assessor. | Week 26

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Dermatology, Redwood City, California
  - Mission Dermatology, Santa Margarita, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Massachusetts, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No